CLINICAL TRIAL: NCT03304782
Title: Quantitative Activity Levels and Gestational Age at Delivery: A Prospective Cohort Study Among Nulliparous Women
Brief Title: Fitbit Activity Tracker to Predict Risk of Preterm Birth
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Cynthia Gyamfi, Principal Investigator, Columbia University
Other Study IDs: AAAR3883
Record Dates: First submitted 2017-09-29; First posted 2017-10-09 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Preterm Birth; Preterm Delivery
Keywords: Preterm Birth; Fitbit; Preterm Delivery
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm birth: Data collected using Fitbit activity tracker from women with delivery prior to 37 weeks gestation
  Interventions: Other: Fitbit activity tracker
- Full-term birth: Data collected using Fitbit activity tracker from women with delivery after 37 weeks gestation
  Interventions: Other: Fitbit activity tracker

INTERVENTIONS:
Other: Fitbit activity tracker — Wearable device that records the number of steps a person takes throughout the day

SUMMARY:
Almost half of all deliveries in the United States are of nulliparous patients. They have been identified as an at-risk population for preterm birth. Historically, the most significant risk factor for preterm birth is a prior history of preterm birth, which cannot be applied to a nulliparous population. Forecasting adverse outcomes in first time moms is difficult to predict and prevent. Historically, physicians have prescribed a restriction in activity level for those at risk for preterm delivery. The utility of this intervention has yet to be prospectively and quantitatively studied. The Fitbit activity tracker is a wearable device that has been extensively used in medical research, in an attempt to quantitatively identify how patient activity levels can improve medical outcomes. The study uses the Fitbit device in nulliparous patients, remotely track their activity levels throughout pregnancy, and assess pregnancy outcomes. Because of the significant and long-standing health disparity in the incidence of preterm delivery, the investigators will use the "Everyday Discrimination Scale", a validated battery of racism and health to see how a patient's stress related to perceived discrimination may modify the risk of preterm delivery.

DETAILED DESCRIPTION:
Preterm birth (PTB) remains one of the leading causes of neonatal morbidity and mortality, with a variety of modifiable and non-modifiable risk factors. In an attempt to prevent PTB, activity restriction is one of the most commonly prescribed interventions in obstetrics, with the idea that decreasing activity will mitigate the risk of a preterm delivery (PTD). However, there has been a lack of evidence in the literature to support this theory. In fact, multiple studies have demonstrated that decreased activity levels have decreased time to delivery in both women with a short cervix, as well as nulliparous patients at increased risk for PTB.

Approximately 40% of deliveries in the United States are nulliparous. For this overwhelming large portion of women, a knowledge gap exists in assessing their risk for PTB. The most powerful risk factor for PTB, a previous PTB, is not applicable to this cohort of women. The precise etiology of PTB in nulliparous women remains unknown but factors found to be associated have included health behaviors , as well as being part of disadvantaged populations. Studies have demonstrated a significant racial disparity in PTB, contributing to the disproportionally worse fetal outcomes in minority populations. Institutional racism, reported stress levels and discrimination have all been identified as risk factors for PTB.

Interventions to prevent PTB have thus far found to be ineffective, and therein likes an opportunity to identify risk factors in this largely unstudied population and create measures, focusing on behavior modification and acknowledging related risks of health disparities to impact maternal and neonatal outcomes.

Currently there are no published prospective studies using quantitative measures to evaluate physical activity in relation to gestational age at delivery. Based on a cohort design, our objective is to use a Fitbit activity tracking device, and assess nulliparous patients. Our hypothesis is that higher physical activity measured in steps per day will be associated with a later gestational age at delivery.

Each participant will be given a Fitbit, complementary of participating in the study. Women will be instructed to wear the Fitbit to measure physical activity throughout the duration of the entire pregnancy, 24 hours a day. The Fitbit has been shown to be valid measure of steps under laboratory conditions. Also, the Fitbit provides estimates of "sedentary", "light", "fairly active" and "very active" minutes as daily accumulated totals. All data from the Fitbit device will be acquired using the Fitabase software system. Fitabase is a research software platform that collects data from devices remotely in near real time as devices sync and update to the Fitabase dashboard. It creates spreadsheet exports of reported data, which can be retrieved remotely by investigators. Fitabase stores the data collected in high security data centers, and only permitted research personnel can access the data.

Upon enrollment in the study, researchers will administer the Fitbit device to each study participant. Researchers will register participants with the Fitabase software system, giving them a unique anonymous patient identifier, which will link each patient and their Fitbit to the Fitabase software system. User accounts will be created by the enrolling researcher for each participant account authorizing access to the Fitbit data for study personnel only. The data collected from the Fitbit is continuously uploaded remotely from the wearable device to the Fitabase software; new information is uploaded every 20 minutes. The device only holds a total of 7 days of patient activity information, so the participant will be required to sync their device to the software system every 7 days. This is done by an app, which is downloaded on the participants' phone at the enrollment of the study. Of note, Fitbit data (ie: steps, activity monitoring) will be blinded to the participants; the Fitbit device has no visible monitoring screen. Research assistants will monitor compliance of participants to syncing their Fitbit and will be sent an email reminder if they do not sync the Fitbit within the last five days. Days with '0' minutes of registered activity will be considered non-valid and set to missing.

ELIGIBILITY:
Inclusion Criteria:

* Documented single viable intrauterine pregnancy at the time of enrollment
* Nulliparous women
* At least 18 years of age
* Access to a smartphone or computer

Exclusion Criteria:

* Known or suspected major congenital anomalies or aneuploidy
* Fetal demise
* Multiple gestation
* Known maternal medical complications (increasing patient risk for indicated (planned) preterm delivery:

  * Pre-gestational diabetes White's Class D or worse
  * Cancer (undergoing treatment)
  * Current hyperthyroidism if not adequately controlled
  * Renal disease with altered renal function (serum creatinine > 1.5)
  * Systemic lupus, scleroderma, polymyalgia rheumatica
  * Active liver disease (acute hepatitis, chronic active hepatitis, persistently abnormal liver enzymes)
  * Platelet or red blood cell disorder
  * Chronic pulmonary disease (aside from asthma)
  * Structural, functional or ischemic heart disease. Neither mitral valve prolapse nor paroxysmal supraventricular tachycardia are considered exclusions.
  * Known HIV positive with viral load greater than 1,000 copies/ml or cluster of differentiation 4 (CD4) count less than 350/mm3
  * Current or planned cerclage
  * Planned delivery prior to 37 weeks
  * Planned delivery at a non-participating hospital
* Patients who do not have regular access to a smart phone or computer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are having their first baby, and have a low risk pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Difference in number of steps | Duration of pregnancy (< 9months)
  The difference in steps per day between women that deliver preterm versus those that deliver at term will be analyzed.

SECONDARY OUTCOMES:
Average number of steps for those women who deliver prior to 37 weeks gestation | Duration of pregnancy (< 9months)
  Average number of steps for those women who deliver prior to 37 weeks gestation
Average number of steps for those women who delivery prior to 34 weeks gestation | Duration of pregnancy (< 9months)
  Average number of steps for those women who delivery prior to 34 weeks gestation
Change in steps per week | Duration of pregnancy (< 9months)
  Change in steps per week over each trimester
Number of triage visits | Duration of pregnancy (< 9months)
  Number of triage visits for threatened preterm labor
Number of inpatient hospitalizations | Duration of pregnancy (< 9months)
  Number of inpatient hospitalizations for threatened preterm labor
Incidence of adverse maternal outcomes | Duration of pregnancy (<9months)
  Incidence of adverse maternal outcomes including pre-eclampsia, diabetes
Incidence of adverse fetal outcomes | Duration of pregnancy (<9months)
  Incidence of adverse fetal outcomes including Intrauterine growth restriction (IUGR), oligohydramnios, placental abruption
Incidence of cesarean section | Duration of pregnancy (< 9months)
  Incidence of cesarean section
Pregnancy physical activity questionnaire (PPAQ) | Duration of pregnancy (< 9months)
  The PPAQ is a validated, self-administered questionnaire that takes on average 10-15 minutes to complete, and has been used to assess the current physical activity levels of pregnant women. This questionnaire is composed of 32 questions, grouped into different types of activities. an estimated average metabolic equivalent (MET-hr/wk) value will be calculated. Clinical practice guidelines have shown that achieving 8.5 MET-hr/wk is associated with healthy gestational weight gain (GWG).
Perceived Stress Scale (PSS) | Duration of pregnancy (< 9months)
  The PSS is a classic stress assessment instrument. For each question, the answers are ranked as follows: 0 - never, 1 - almost never, 2 - sometimes, 3 - fairly often, 4 - very often. A calculated total score can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 - low stress; 14-26 - moderate stress; 27-40 - high perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Gyamfi, M.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Booker WA, Ekpe EE, Handal-Orefice RC, Zhang Y, Cande A, Gyamfi-Bannerman C, Nieto V. Quantitative activity levels and gestational age at delivery: a prospective cohort study among nulliparous women. Am J Obstet Gynecol MFM. 2022 Jan;4(1):100503. doi: 10.1016/j.ajogmf.2021.100503. Epub 2021 Oct 17. PMID 34666197